CLINICAL TRIAL: NCT05578690
Title: Healthy Lifestyle Before and During Pregnancy to Prevent Childhood Obesity. A Randomized, Parallel Group, Tailored Multifactorial Lifestyle Intervention Trial Among Women With Overweight or Obesity Seeking Pregnancy - the PRE-STORK Trial
Brief Title: Healthy Lifestyle Before and During Pregnancy to Prevent Childhood Obesity - the PRE-STORK-trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-22011403
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obesity; Pregnancy Related
Keywords: Diet; Exercise; Mentors
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: The trial is a randomised, parallel-group, intervention study comparing a tailored, intensive, multifactorial lifestyle intervention before and during pregnancy in women with overweight or obesity with standard of care.
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis of the primary outcome will be blinded to the assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle group (Experimental): A tailored multifactorial lifestyle intervention consisting of diet, exercise and mentorship in women with overweight or obesity to obtain a healthy lifestyle before and during pregnancy.
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Mentorship
- Standard of care group (No Intervention): The standard of care group will receive no active intervention but are encouraged to seek any possible guidance from the general practitioner for management of pre-pregnancy obesity according to current guidelines.

INTERVENTIONS:
Behavioral: Diet — An initial 8 weeks of low-calorie diet including meal replacements (total of 800 kcal/day) will be initiated with the objective to lose at least 10% of initial body weight. From week 8 until week 12, an individual food-reintroduction plan will take place with partial meal product substitution. At week 12 and until pregnancy dieticians will ensure sustained compliance with diet aligned with the general recommendations for women seeking pregnancy (low-fat diet, rich in protein and carbohydrates and in some individuals slightly carbohydrate-reduced diet (prediabetes or family disposition to diabetes) with focus on carbohydrate quality (more fiber and whole grain). Consultations with a dietician for mapping diet and eating patterns and regular follow-up with a dietitian to maintain diet changes and modify diets if needed.
  Arms: Lifestyle group
Behavioral: Exercise — After an initial 8-week ramp-up phase (during the initial low-calorie diet), the women will be encouraged to attend supervised exercise sessions on the study location (combination of vigorous-intensity, interval-based indoor cycling, and circuit training) twice weekly and to perform additional moderate-to vigorous-intensity exercise to obtain at least 150 min per week of moderate-intensity or 75 min per week of vigorous-intensity physical activity or a combination. The plan will include individual exercise and/or group exercise. Exercise watches with heart-rate monitors will be worn at each exercise session to determine whether the requirement regarding weekly time spent at moderate or vigorous intensity will be met. Regular follow-up with the women to maintain exercise changes and modify the exercise plan if needed.
  Arms: Lifestyle group
Behavioral: Mentorship — Women are offered an individualized plan to successfully fulfil the multifactorial lifestyle intervention and the women will be offered both individual and/or group sessions with a mentor. After 8 weeks of the intervention, the women will be invited to another meeting where the choice of mentor will be evaluated, and the women will be offered to join a "pre-parents-group". Group sessions will include conversational sessions, cooking classes and exercise classes with focus on changing lifestyle and maintaining a healthy lifestyle change. At the time of pregnancy groups will be reconsidered and the women will be offered participation in "pregnancy-groups".
  Arms: Lifestyle group

SUMMARY:
Introduction: The prevalence of childhood overweight and obesity has risen from just 4% in 1975 to more than 18% in 2016. Little is known about adiposity of the infant, but it positively associates to the mother's BMI. Globally, the prevalence of overweight has tripled since 1975 and is now affecting one of three Danish women at the time of pregnancy. However, despite increasing awareness of obesity and accumulating evidence of its health consequences limited effect of intervention in childhood obesity exists. Maternal obesity before conception, an excessive increase in body weight during pregnancy and physical inactivity are some of the risk factors suspected of infant adiposity. Lifestyle interventions during pregnancy have shown limited or no effect in the offspring. Therefore, renewed effort to improve the prevention of childhood obesity is warranted.

Methods and analysis: This is a randomized, parallel group, tailored, multifactorial lifestyle intervention trial in women (age 18 to 38 years) with overweight or obesity (BMI 27 to 42 kg/m2) seeking pregnancy. The women are randomized 1:1 to either the lifestyle or standard of care group. The lifestyle intervention is initiated prior to pregnancy. The lifestyle intervention is set off with a low-calorie diet for 8 weeks and throughout the intervention period (prior to and during pregnancy) participants follow an intervention containing exercise according to the World Health Organization guidelines, healthy diet and mentorship to maintain healthy weight before and during pregnancy.The primary outcome is the difference in neonatal adiposity measured at birth. Finally, a child and family cohort will be established to follow the children throughout childhood for healthy weight development. The study will provide evidence of effects from pre-conception-initiated intervention and have the potential to improve health and quality of life for children.

Ethics and dissemination: The trial has been approved by the ethical committee of the Capital Region of Denmark (H-22011403) The trial will be conducted in agreement with the Declaration of Helsinki and monitored to follow the guidelines for good clinical practice. Results will be submitted for publication in international peer-reviewed scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Having overweight or obesity (BMI 25-44 kg/m2)
* Age 18-34 years (no previous pregnancy) or 18-40 years (previous pregnant >16 weeks)
* Planning a pregnancy within the next year
* Willingness to lose at least 10% of initial body weight before pregnancy and be physically able to adhere to WHO physical activity recommendations when entering the study
* Willing to postpone pregnancy until at least 6 months after randomization
* Planning antenatal care and delivery at either Herlev Hospital or Odense University Hospital
* Danish or English speaking

Exclusion Criteria:

* Diabetes (fasting plasma glucose (FPG) >7 mmol/l and HbA1c ≥48 mmol/mol)
* Previous gestational diabetes mellitus (GDM) treated with insulin during pregnancy
* Polycystic ovary syndrome (PCOS) treated with metformin
* Treatment with medication which significantly affect glucose metabolism, appetite, or energy balance
* The use of medications that cause clinically significant weight gain or loss
* Habitual abortion (more than 3 abortions in a row)
* Known infertility (defined as fertility treatment and/or no obtained conception with the same partner after trying >12 months)
* Previous bariatric surgery
* Significant psychiatric disorders
* Uncontrolled/severe medical issues including cardiovascular, pulmonary, rheumatologic, hematologic, oncologic, infectious, or endocrine disease
* Regular exercise training at high intensity (e.g., spinning) >3 hours per week
* Known eating disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women who have overweight or obesity seeking pregnancy (with no known fertility problems) are eligible if having a BMI between 25-44 kg/m2 and in the age range of 18-40 years.
Enrollment: 360 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Neonatal adiposity | Assessed at birth or up to 72 hours postpartum.
  Total fat mass (in gram) assessed by air displacement plethysmography (PEA POD).

SECONDARY OUTCOMES:
Foetal and infant body weight | Assessed during pregnancy (week 18-21, 24-28 and 34), at birth and 3 months after birth.
  During pregnancy foetal body weight is determined by ultrasonographic method and infant body weight is measured on a scale.
Foetal and infant abdominal circumference | Assessed during pregnancy (week 18-21, 24-28 and 34), at birth and 3 months after birth.
  During pregnancy abdominal circumference is determined by ultrasonographic method and infants are measured to the nearest 1.0 cm.
Foetal and infant femur length | Assessed during pregnancy (week 18-21, 24-28 and 34), at birth and 3 months after birth.
  During pregnancy femur length is determined by ultrasonographic method and infants are measured to the nearest 1.0 cm.
Foetal and infant head circumference | Assessed during pregnancy (week 18-21, 24-28 and 34), at birth and 3 months after birth.
  During pregnancy head circumference is calculated by biparietal diameter and occiput-frontal diameter by ultrasonographic method and infants are measured to the nearest 1.0 cm.
Placenta function (during pregnancy) | Assessed during pregnancy (week 34).
  Measured by the represented amount of amniotic fluid, cerebral media and umbilical artery doppler flow of the foetus.
Neonatal body mass index (BMI) z-score | Assessed at birth.
  Body mass index (BMI) is body weight relative to height (kg/m^2) and BMI z-score is called BMI standard deviation (s.d.) scores and is a measure of relative weight adjusted for child age and sex.
Neonatal body composition (fat percent) | Assessed at birth.
  Measured by air displacement plethysmography (PEA POD).
Neonatal body composition (fat free mass) | Assessed at birth.
  Measured by air displacement plethysmography (PEA POD) and lean mass is also based on this assessment.
Gestational age | Assessed at birth.
  The gestational age is registered when giving birth.
Weight for gestational age | Assessed at birth.
  Measured as percent of normal weight related to gestational age.
Large for gestational age (LGA) | Assessed at birth.
  Assessed as the proportions of infants being born LGA
Small for gestational age (SGA) | Assessed at birth.
  Assessed as the proportions of infants being born SGA.
Apgar score | Assessed at birth.
  Assessed as the proportions of infants born with Apgar score <7.
Placenta function (birth) | Assessed at birth.
  Assessed by the weight of the placenta (in gram).
Faeces (infant) | Assessed at birth and 3 months after birth.
  Changes in faecal microbiota composition.
Infant body composition (fat mass, fat free mass) PEA POD | Assessed 3 months after birth
  Body composition (fat mass (g), and fat free mass (g)) is assessed by air displacement plethysmography (PEA POD).
Infant body composition (fat percent) PEA POD | Assessed 3 months after birth
  Body composition (fat percent (%) ) is assessed by air displacement plethysmography (PEA POD).
Infant body composition (fat mass, fat free mass) dual energy x-ray absorptiometry. | Assessed 3 months after birth.
  Body composition (fat mass (g) and fat free mass (g)) is assessed by dual energy x-ray absorptiometry scans.
Infant body composition (fat percent) dual energy x-ray absorptiometry. | Assessed 3 months after birth.
  Body composition (fat percent (%)) is assessed by dual energy x-ray absorptiometry scans.
Infant BMI z-score | Assessed 3 months after birth.
  Body mass index (BMI) is body weight relative to height (kg/m^2) and BMI z-score is called BMI standard deviation (s.d.) scores and is a measure of relative weight adjusted for child age and sex.
Weight loss (women) | Assessed up to 2 years.
  Assessed as the proportion of women who achieve a weight loss of ≥10% at time of pregnancy (or two years after randomisation without achieving pregnancy)
Pregnancy (women) | Assessed up to 2 years.
  Assessed as the proportion of women without obtaining pregnancy or live-born offspring within a period of two years.
Glucose tolerance (OGTT) | Assessed during pregnancy (week 24-28)
  Maximum observed glucose concentration, time to maximum observed glucose concentration and baseline-subtracted area under the plasma glucose concentration time curve (0-120 min), and two-hour plasma glucose concentration are assessed during a 75 gram oral glucose tolerance test.
Insulin resistance (fasting insulin) | Assessed during pregnancy (week 24-28).
  Fasting insulin concentration is assessed prior to a 75 gram oral glucose tolerance test.
Insulin resistance (OGTT) | Assessed during pregnancy (week 24-28).
  Area under the insulin concentration time curve (0-60 min), area under the insulin concentration time curve (0-120 min), maximum observed insulin concentration, time to maximum observed insulin concentration, baseline-subtracted area under the insulin concentration time curve (0-60 min) and baseline-subtracted area under the insulin concentration time curve (0-120 min), Matsuda index and homeostasis model assessment-insulin resistance (HOMA-IR) are assessed during a 75 gram oral glucose tolerance test.
Hormonal response - glucagon (OGTT) | Assessed during pregnancy (week 24-28).
  Glucagon assessed during a 75 gram oral glucose tolerance test.
Hormonal response - GLP-1 (OGTT) | Assessed during pregnancy (week 24-28).
  Glucagon-like peptide-1 (GLP-1) assessed during a 75 gram oral glucose tolerance test.
Hormonal response - PYY (OGTT) | Assessed during pregnancy (week 24-28).
  Peptide tyrosine tyrosine (PYY) assessed during a 75 gram oral glucose tolerance test.
Hormonal response - GIP (OGTT) | Assessed during pregnancy (week 24-28).
  Gastric inhibitory peptide (GIP) assessed during a 75 gram oral glucose tolerance test.
Hormonal response - ghrelin (OGTT) | Assessed during pregnancy (week 24-28).
  Ghrelin assessed during a 75 gram oral glucose tolerance test.
Glycaemic variability (CGM and OGTT) | Assessed during pregnancy (week 24-28).
  Measured by 10-day coefficient of variance (CV) of glucose levels measured by continous glucose monitoring (CGM) and during a 75 gram oral glucose tolerance test.
BMI (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months), during pregnancy (week 11-14, 18-21, 24-28 and 34) and 3 months after giving birth.
  Calculated as weight (kg) divided by height(m)^2.
Body weight (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months), during pregnancy (week 11-14, 18-21, 24-28, 34, 38 and at delivery) and 3 months after giving birth.
  Measured by scale to nearest 0.1 kg
Height (women) | Assessed prior to pregnancy (baseline).
  Measured to the nearest 0.5 cm.
Body composition (fat percent and muscle mass percent) (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months), during pregnancy (week 11-14, 18-21, 24-28 and 34) and 3 months after giving birth.
  Body composition measured by Dual-energy X-ray absorptiometry scans prior to and after pregnancy. During pregnancy measured by bioelectrical impedance analysis.
Bone density (T-score) (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months) and 3 months after giving birth.
  Bone density is measured by Dual-energy X-ray absorptiometry scans prior to and after pregnancy. During pregnancy measured by bioelectrical impedance analysis.
Resting heart rate (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months), during pregnancy (week 11-14, 18-21, 24-28 and 34) and 3 months after giving birth.
  After resting for a minimum of 10 minutes heart rate measured 3 times with 2 min in between each measurement.
Blood pressure (women) | Assessed prior to pregnancy (baseline, 6 months, 12 months), during pregnancy (week 11-14, 18-21, 24-28 and 34) and 3 months after giving birth.
  After resting for a minimum of 10 minutes systolic and diastolic blood pressure is measured 3 times with 2 min in between each measurement.
Fasting plasma glucose (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Fasting plasma glucose is measured by blood sampling after an overnight of fasting.
HbA1c (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  HbA1c is measured by blood sampling after an overnight of fasting.
Lipid profile - cholesterol (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Cholesterol is measured by blood sampling after an overnight of fasting.
Lipid profile - HDL (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  High-density lipoprotein (HDL) is measured by blood sampling after an overnight of fasting.
Lipid profile - LDL (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Low-density lipoprotein (LDL) is measured by blood sampling after an overnight of fasting.
Lipid profile - VLDL (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Very-low-density lipoprotein (VLDL) is measured by blood sampling after an overnight of fasting.
Lipid profile - TG (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Triglycerides is measured by blood sampling after an overnight of fasting.
Lipid profile - ApoA/ApoB ratio (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Apolipoprotein B/apolipoprotein A1 ratio assessed by blood sampling after an overnight of fasting.
Liver function - liver fat (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Liver function by Fibro-Scan (a proxy for liver fibrosis) measured by Fibro-Scan (UL-based elastography) and liver fat is measured by the controlled attenuation parameter score in decibel per meter.
Liver function - liver stiffness (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Liver function by Fibro-Scan (a proxy for liver fibrosis) is measured by Fibro-Scan (UL-based elastography) and liver stiffness is measured by shear wave velocity in kilopascal.
Food preference (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Food preference is measured using the Steno Biometric Food Preference Task after an overnight of fasting.
Bone homeostasis - CTX (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Pharmacodynamic endpoints for bone homeostasis derived from bone turnover markers carboxy-terminal collagen crosslinks (CTX) as a marker for bone resorption after an overnight of fasting.
Bone homeostasis - P1NP (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Pharmacodynamic endpoints for bone homeostasis derived from bone turnover markers type 1 amino-terminal pro-peptide (P1NP) as a marker for bone formation after an overnight of fasting.
Bone homeostasis - OC (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Pharmacodynamic endpoints for bone homeostasis derived from bone turnover markers osteocalcin (OC) as a marker of bone formation after an overnight of fasting.
Inflammatory markers - hs-CRP (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28), at delivery and 3 months after giving birth.
  High-sensitivity C-reactive protein (hs-CRP) is measured by blood sampling after an overnight of fasting.
Inflammatory markers - TNFa (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Tumour necrosis factor-α (TNF-α) is measured by blood sampling after an overnight of fasting.
Inflammatory markers - IL-6 (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Interleukin-6 (IL-6) is measured by blood sampling after an overnight of fasting.
Inflammatory markers - LBP (women) | Assessed prior to pregnancy (baseline and 6 months) during pregnancy (week 24-28) and 3 months after giving birth.
  Lipopolysaccharide-binding protein (LBP) is measured by blood sampling after an overnight of fasting.
Waist and hip circumference (women) | Assessed prior to pregnancy (baseline, 8 weeks, 6 months, 12 months and 18 months) and 3 months after giving birth.
  Waist and hip circumference is measured to the nearest 0.1 cm.
Resting energy expenditure (women) | Assessed prior to pregnancy (baseline, 6 months, and three months after giving birth)
  Resting energy expenditure is meaured using indirect calorimetry.
Exercise capacity (women) | Assessed prior to pregnancy (baseline, 6 months, and three months after giving birth)
  Exercise capacity is measured by maximal exercise test with direct measurement of maximal oxygen consumption.
Prediabetes (women) | Assessed prior to pregnancy (6 months from baseline)
  Assessed as the proportion of women with prediabetes.
Gestational diabetes (women) | Assessed during pregnancy (week 10 to 40)
  Assessed as the proportion of women diagnosed with gestational diabetes according to the Danish guidelines
Exercise capacity (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 24-28), and three months after giving birth)
  Exercise capacity is measured indirectly with the decive Seismofit® which estimates the maximal oxygen consumption by a 3-minute test during rest using seismocardiography.
Daily physical activity, sedentary time and sleep (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 24-28), and 3 months after giving birth)
  Daily physical activity, sedentary time and sleep are measured with an 3-axis accelerometer (AX3, Axivity) for seven consecutive days. Two devices are placed on lower back and the thigh, respectively.
Duration and intensity of physical exercise (women in the intervention group) | The women in the intervention group will be wearing the watch 24 hour/day from baseline to 3 months after giving birth.
  Physical exercise duration and intensity, daily physical and sleep are measured in the intervention group by a activity watch.
Hypertensive disorders in pregnancy | Will be obtained from electronical medical records from gestational week 20 until 48 hours post partum
  Defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHG
Pre-eclampsia | Will be obtained from electronical medical records from gestational week 20 until 48 hours post partum
  If hypertension occurs during pregnancy, information on the findings below will be obtained:
  i. proteinuria > 0,3 gram/liter ii. Thrombocytopenia (< 100x109/l) iii. Renal insufficiency (serum creatinine > 100 mmol/l) iv. Impaired liver function (elevated transaminases to twice the normal concentration) v. Pulmonary edema vi. Cerebral or visual symptoms vii. Utero-placental dysfunction (SGA corresponding to an ultrasound-estimated weight below -15 %)
Essential hypertension | Will be obtained from electronical medical records prior to pregnancy until gestational week 20.
  Defined as diagnosed hypertension before gestional week 20
Mode of delivery | Assessed at birth
  Destinction between
  * Non-instrumental vaginal delivery
  * Instrumental vaginal delivery
  * Elective caesarean section
  * Emergency caesarean section (grade 1,2 or 3)
Breastfeeding practice | Assessed by individual questionnaire 4 months after giving birth
  Successful breastfeeding 12 weeks after delivery, defined as exclusive breastfeeding (using formula supplements less than once a week)
Brest milk composition | Samples will be collected within 72 hours post partum, and at week 12 after delivery
  Analyses will consist of analysing macronutrient content (protein, fat, carbohydrates, and calories), vitamins and minerals

OTHER OUTCOMES:
Fertility treatment (women) | Assessed up to 2 years.
  Assessed as the proportion of women who initiate fertility treatment during the trial period
Body weight (partner) | Assessed prior to pregnancy of the woman (baseline and 6 months), during pregnancy (week 11-14) and 3 months after birth.
  Body weight is measured using a scale to the nearest 0.1 kg.
Height (partner) | Assessed prior to pregnancy of the woman (baseline)
  Height is measured to the nearest 0.5 cm.
BMI (partner) | Assessed prior to pregnancy of the woman (baseline and 6 months), during pregnancy (week 11-14) and 3 months after birth.
  BMI is calculated as weight (kg) divided by height(m)^2.
Body composition - fat mass and fat free mass (partner) | Assessed prior to pregnancy of the woman (baseline and 6 months), during pregnancy (week 11-14) and 3 months after birth.
  Fat mass (g) and fat free mass (g) are measured by bioelectrical impedance analysis after standardized conditions.
Body composition - fat percent (partner) | Assessed prior to pregnancy of the woman (baseline and 6 months), during pregnancy (week 11-14) and 4 months after birth.
  Fat percent (%) is measured by bioelectrical impedance analysis after standardized conditions.
Blood pressure (partner) | Assessed prior to pregnancy of the woman (baseline and 6 months), during pregnancy (week 11-14) and 3 months after birth.
  After resting for a minimum of 10 minutes systolic and diastolic blood pressure is measured 3 times with 2 min in between each measurement.
Appetite, physical activity and wellbeing (women and partner) | Assessed prior to pregnancy (baseline and 6 months), during pregnancy (week 24-28) and 3 months after birth
  Appetite sensation, daily physical activity level and wellbeing based on questionnaires.
Sleep (women and partner) | Assessed prior to pregnancy (baseline and 6 months), during pregnancy (week 24-28) and 3 months after birth.
  Sleep patterns based on questionnaires.
Self perception of body weight, self-esteem and partner support (women and partner) | Assessed prior to pregnancy (baseline and 6 months), during pregnancy (week 24-28) and 3 months after birth.
  Perception of weight-related stigma and self-esteem, social/partner support on eating habits and exercise based on questionnaires.
Semen quality (partner) | Assessed prior to pregnancy of the woman (baseline) and during pregnancy (week 11-14).
  Quality of semen from the father (meassured as number of sperm cells).
Semen epigenetics (partner) | Assessed prior to pregnancy of the woman (baseline) and during pregnancy (week 11-14).
  Epigenetic profile of sperm cells
Umbilical cord | Assessed at birth.
  Epigenetic profile from umbilical cord blood
Placenta | Assessed at birth.
  Epigenetic profile from placenta biopsies
Epigenetic (women, partner and child) | Assessed at birth.
  Epigenetic profile in peripheral blood mononuclear cells
Faeces (women) | Assessed prior to pregnancy (baseline) and 3 months after birth.
  Changes in faecal microbiota composition,: (what species are present and how many different types of species are present with a sample) using Shannon index.
Obesity related-phenotypes | Assessed at the end of the trial intervention period.
  Associations between parent and child genetics and obesity-related phenotypes.
Complications (delivery) | Assessed at birth.
  Proportion of women who experience complications during delivery (premature delivery, labour induction, vacuum extraction, shoulder dystocia, planned and emergency caesarean section, postpartum haemorrhage and stillbirth).
Neonatal complications (delivery) | Assessed at birth.
  Proportion of children with neonatal complications including (simple and complex) asphyxia (represented by potential of Hydrogen (pH)-values from umbilical cord), hypoglycaemia, jaundice, and admittance to neonatal intensive care
Thrombelastography (TEG) (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 11-14 and 24-28), at birth and 3 months after giving birth.
  TEG is measured by blood sampling after an overnight of fasting
Complications during pregnancy (gestational week 24 - 40) | Assessed during pregnancy (week 24-40) and 3 months post-partum
  Proportion of women who experience complications during pregnancy (gestational week 24 - 40) and post-partum (3 months post partum) (deep vein thrombosis, pulmonary embolism, gestational hypertension, preeclampsia, abortion)
International Normalized Ratio in umbillical cord (child) | Assessed at birth
  International Normalized Ratio (combined measure for coagulation factor II, VII, and X). Blood sampled from umbillical cord at birth.
Haemoglobin (child) | Assessed at birth
  Concentration of haemoglobin is measured by blood sampling from umbillical cord at birth
High-sensitivity C-reactive protein (child) | Assessed at birth
  Concentration of high-sensitivity CRP (hsCRP). Blood sampled from umbillical cord at birth
Liver marker alanine transaminase (child) | Assessed at birth
  Concentration of alanine transaminase. Blood sampled from umbillical cord at birth
Thrombelastography (TEG) (child) | Assessed at birth and 3 months after birth
  TEG is measured by blood sampled from umbillical cord at birth and from vein puncture three months after birth
Concentration of endothelial marker thrombomodulin (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 11-14 and 24-28), at delivery and three months after giving birth.
  Concentration of the endothelial marker thrombomodulin, is measured by blood sampling after an overnight of fasting.
Coagulation function (Child) | Measured at birth.
  Activated partial thromboplastin time (seconds)(APTT). Blood sampled from umbillical cord at birth.
Coagulation ratio (Child) | Measured at birth.
  International normalised ratio (INR) of time (seconds). Blood sampled from umbillical cord at birth.
Liver marker bilirubin (Child) | Measured at birth
  Concentration of bilirubin. Blood sampled from umbillical cord at birth
Liver marker albumin (Child) | Measured at birth
  Concentration of albumin. Blood sampled from umbillical cord at birth
Endothelial marker Syndecan-1 (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 11-14 and 24-28), at delivery and three months after giving birth.
  Concentration of syndecan-1 is measured by blood sampling after an overnight of fasting.
Endothelial marker PECAM-1 (women) | Assessed prior to pregnancy (baseline, 6 months), during pregnancy (week 11-14 and 24-28), at delivery and three months after giving birth.
  Concentration of platelet endothelial cell adhesion molecule 1 (PECAM-1) is measured by blood sampling after an overnight of fasting.
Self-perception of the severity of pregnancy-related nausea and vomiting (women) | Assessed once weekly from registration of pregnancy (week 5-10) until delivery (week 40).
  The severity of pregnancy-related nausea and vomiting is meas-ured based on the questionnaire Pregnancy-Unique Quantification of Emesis and Nausea (PUQE)
Planned obstetric consultations | Will be obtained from electronical medical records from gestational week 20 until 48 hours post partum
  Number of planned obstetric consultations after gestational week 20
Obstetric emergency consultations | Will be obtained from electronical medical records from gestational week 20 until 48 hours post partum
  Number of obstetric emergency consultations after gestational week 20
Urinary tract infections during pregnancy | Will be obtained from electronical medical records from gestational week 20 until 48 hours post partum
  Number of diagnosed urinary tract infections during pregnancy
Vaginal bleeding in pregnancy | Will be obtained from electronical medical records from gestational week 20 until birth
  Number of admissions with vaginal bleeding episodes after gestational week 20
Premature contractions | Will be obtained from electronical medical records from gestational week 20 until birth
  Admissions with premature contractions before gestational week 34
Shortened cervix | Will be obtained from electronical medical records from gestational week 20 until birth
  Admissions with shortened cervix less than 20 mm before gestational week 34
Preterm delivery | Will be obtained from electronical medical records from gestational week 20 until birth
  Defined as delivery before gestational week 34
Induction of labour | Will be obtained from electronical medical records from gestational week 20 until birth
  Induction (mechanical or medical) of labour before spontaneous onset of labour
Epidural analgesia | Will be obtained from electronical medical records from admission to the labour ward until birth
  Use of epidural analgesia during birth
Scalp pH sampling | Will be obtained from electronical medical records from admission to the labour ward until birth
  Use of scalp pH sampling during birth
Oxytocin stimulation | Will be obtained from electronical medical records from admission to the labour ward until birth
  Use of Oxytocin stimulation in active labour
Perineal lacerations | Will be obtained from electronical medical records from the time of birth until 48 hours post partum
  Perineal lacerations, destinction between 1st, 2nd, 3rd, and 4th degree
Post-partum haemorrhage | Will be obtained from electronical medical records from the time of birth until 48 hours post partum
  Post-partum haemorrhage in mL
Admission and re-submission after delivery | Will be obtained from electronical medical records from the time of birth until 12 weeks post partum
  Length of admission and re-submission after delivery
Anaemia during and after pregnancy | Will be obtained from electronical medical records from gestational week 20 until 12 weeks post partum
  Defined as haemoglobin less than 5.0 mmol/l
Mastitis | Will be obtained from electronical medical records from the time of birth until 12 weeks post partum
  Diagnosed mastitis
Endometritis | Will be obtained from electronical medical records from the time of birth until 12 weeks post partum
  Diagnosed Endometritis
Hospital admissions | Will be obtained from electronical medical records from gestational week 20 until 12 weeks post partum
  Number of and total length of hospital admissions
Mood and depressions | Will be assessed by individual questionnaire 4 months after giving birth
  Mood and depressions Edinburgh Postnatal Depression Scale 16 weeks after delivery
Quality of life (SF-36) | Will be assessed by individual questionnaire 4 months after giving birth
  Quality of life (SF-36) 16 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, Professor, Principal Investigator — Steno Diabetes Center Copenhagen; Louise G. Grunnet, PhD, Principal Investigator — Steno Diabetes Center Copenhagen; Signe Torekov, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request. The dataset contains protected health information and will not be available online. Study results will be available by contacting the corresponding author. A proposal must be submitted to the PRE-STORK steering committee. If approved, data will be available.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Kornerup N, Danielsen JH, Sahl RE, Pico ML, Johansen MY, Knop FK, Bonnelykke K, Bergholt T, Kelstrup L, Foghsgaard S, Ghauri N, Gronlund E, Lund L, Vinter CA, Lyng Forman J, Barres R, Kragelund Nielsen K, Andersen A, Torekov SS, Groth Grunnet L, Vilsboll T. Healthy lifestyle before and during pregnancy to prevent childhood obesity: study protocol for a parallel group randomised trial - the PRE-STORK trial. BMJ Open. 2025 Jan 25;15(1):e087895. doi: 10.1136/bmjopen-2024-087895. PMID 39863406